CLINICAL TRIAL: NCT06591299
Title: Combining Aspirin With Cilostazol or Clopidogrel in Minor Stroke or TIA, a Randomized Controlled Trial
Brief Title: Combining Aspirin With Cilostazol or Clopidogrel in Minor Stroke or TIA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Mohamed G. zeinhom, MD, principal investigator, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23098816714
Record Dates: First submitted 2024-09-08; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Ischemic Stroke
Keywords: cilostazol; clopidogrel; minor stroke; Egypt
MeSH Terms: conditions — Ischemic Stroke | interventions — Cilostazol; Clopidogrel

STUDY DESIGN:
Intervention Model Description: The investigators will conduct our single-blinded randomized controlled trial, which will contain two arms; the clopidogrel arm will receive (a 300 mg loading dose during the first 24 hours of stroke onset, followed by 75 mg daily from the 2nd to the 90th day). The cilostazol arm will receive (a 200mg loading dose during the first 24 hours of stroke onset, followed by 100 mg twice daily from the 2nd to the 90th day). both groups received open-labelloading dose 300 mg aspirin and continued on open-label aspirin 75 mg daily
Who Masked: Investigator, Outcomes Assessor
Masking Description: An independent statistician generated a blocked randomization sequence using computer-generated random numbers; in a one-to-one ratio, participants were randomly assigned to receive loading doses of clopidogrel and aspirin or cilostazol and aspirin by a specially trained and qualified nurse. We prepared Sequentially numbered opaque sealed envelopes and 870 labels for each drug labeled Drug A or B. According to the randomization chart, put them into envelopes numbered 1 to 870. Envelopes were attached to the patient's files. Patients were recruited sequentially and were given enrollment numbers starting from 1, which were mentioned in their files. Files with the same number as the patient enrolment number were opened, and the patients were assigned to receive drugs A or B. Drug A included clopidogrel, and Drug B included cilostazol. Both groups received an open-label loading dose of 300 mg of aspirin and continued on aspirin 75 mg daily.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- cilostazol and aspirin (Active Comparator): The cilostazol arm will receive (a 200 mg loading dose of cilostazol during the first 24 hours of stroke onset, followed by 100 mg twice daily from the 2nd day to the 90th day) and an open-label loading 300 mg aspirin, followed by a maintenance dose of 75 mg aspirin.
  Interventions: Drug: Cilostazol 100 MG
- clopidogrel and aspirin (Active Comparator): The clopidogrel arm will receive (a 300 mg loading dose of clopidogrel during the first 24 hours of stroke onset, followed by 75 mg once daily from the 2nd day to the 90th day) and open-label loading 300 mg aspirin, followed by a maintenance dose of 75 mg aspirin.
  Interventions: Drug: Clopidogrel 75mg

INTERVENTIONS:
Drug: Cilostazol 100 MG — Efficacy and safety of 200 mg cilostazol followed by 100 mg twice daily for three months and loading 300 mg aspirin and 75 mg aspirin maintenance will be assessed through NIHSS, mRS, duration of hospital stay, new ischemic stroke, and possible adverse effects,
  Other Names: group A
  Arms: cilostazol and aspirin
Drug: Clopidogrel 75mg — Efficacy and safety of 300 mg clopidogrel followed by 75mg once daily for three months and loading 300 mg aspirin and 75 mg aspirin maintenance will be assessed through NIHSS, mRS, duration of hospital stay, new ischemic stroke, and possible adverse effects,
  Other Names: group B
  Arms: clopidogrel and aspirin

SUMMARY:
Along with the current clinical trial, the efficacy and safety of a 300 mg loading dose of clopidogrel administered within 24 hours of the first-ever minor stroke or TIA compared to 200 mg cilostazol were assessed through NIHSS, mRS, and possible adverse effects

DETAILED DESCRIPTION:
The investigators conducted a single-blinded randomized controlled trial after the ethics committee of the faculty of medicine at Kafr el-Sheik University approved it.

The investigators got written informed consent from all eligible patients or their first order of kin before randomization.

The study will be composed of 2 arms clopidogrel arm, which consisted of 435 patients who received a 300 mg loading dose followed by 75 mg once daily from the 2nd to the 90th day), and the cilostazol arm, consisting of 435 patients who received (a 200 mg loading dose during the first 24 hours of stroke onset followed by 100 mg twice daily from the 2nd day to the 90th day),

Study Procedures:

Every patient in our study will undergo:

clinical workup: History, clinical assessment & NIHSS were recorded on admission, day 7, and the Modified Rankin Scale as a follow-up after one week and 3 months.

Detection of Risk Factors & Profiles:

Echocardiography TTE: in indicated patients ECG Monitoring: daily ECG monitoring will be performed in indicated patients. 3- Carotid Duplex: carotid duplex in indicated patients.

4- ESR & Lipid Profile& liver functions: All will be tested routinely for all patients.

Imaging Follow-UP Non-contrast CT brain on admission Day 2 MRI: after 2 days of admission, all the patients in this study will have a brain MRI (stroke protocol; T1W, T2W, FLAIR, DWI, T2 Echo Gradient, MRA of all intra-cerebral vessels).

CT brain: Any patient with unexplained clinical deterioration at any time throughout his/her hospital stay will be urgently imaged by CT.

Primary End Point:

The primary efficacy outcome was the rate of new stroke at 90 days, and the primary safety outcome was the rate of drug hemorrhagic complications using the PLATO bleeding definition.

• Secondary End Point: The secondary efficacy outcomes were to evaluate the rates of patients who achieved a significant reduction in NIHSS (decrease of four points or more) at the seventh day or discharge compared to baseline, the rates of a favorable outcome with (mRS = 0-2) after one week and after 90 days in a face-to-face interview in the outpatient clinic, rates of a composite of recurrent stroke, myocardial infarction and death due to vascular events after 90 days of follow-up, while the secondary safety outcome was the rate of treatment-related adverse effects assessed by a follow-up questionnaire

ELIGIBILITY:
Inclusion Criteria:

* the investigators included both genders with eligible ages ranging between 18-75 years, with the first-ever presentation with minor ischemic stroke or TIA who received antiplatelet treatment within the first 24 hours of the onset of ischemic stroke. Patients are not eligible for rt-PA treatment

Exclusion Criteria:

The investigators excluded patients who had not been followed up on for 90 days after enrollment, those with NIHSS < 5 or who had rapidly resolving symptoms before imaging results, and patients with a known history of persistent or recurrent CNS pathology (e.g., epilepsy, meningioma, multiple sclerosis, history of head trauma with a residual neurological deficit).

The investigators excluded patients who had clinical seizures at the onset of their stroke, as well as those who had symptoms of any major organ failure, active malignancies, or an acute myocardial infarction within the previous six weeks, and those who were on warfarin, regular ticagrelor during the week before admission, or chemotherapy within the previous year.

The investigators excluded patients with active peptic ulcers, GIT surgery, bleeding history within the last year, and those with a history of major surgery within the last three months.

The investigators ruled out of our trial patients who had a known allergy to the study drugs and those with INR > 1.4 or P.T. >18 or blood glucose level < 50 or > 400 mg/DL or blood pressure < 90/60 or > 185/110 mmHg on admission or Platelets < 100,000.

The investigators excluded pregnant and lactating patients and those with stroke due to venous thrombosis and stroke following cardiac arrest or profuse hypotension ineligible for our trial.

Patients with contraindications to the study drugs were excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 870 (Estimated)
Dates: Start 2022-04-15 (Actual); Primary Completion 2024-09-15 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
rate of new stroke | 90 days
  Rates of new stroke occur within three months of treatment. The investigators will perform follow-ups of the patient during visits to the outpatient clinic, and brain CT and/ or MRI will be done if there is suspicion of a new stroke.
Rate of drug-related hemorrhagic complications | 90 days
  the rate of drug hemorrhagic complications which was evaluated using the PLATO bleeding definition which classified hemorrhagic complications into three types as follows: Major bleeding which had one or more of the following criteria: fatal bleeding, intracranial, intrapericardial, bleeding associated with reduction of hemoglobin > 3-5 g/dl, bleeding required transfusion of two to four units whole blood or PRBCs, bleeding produced hypovolemic shock or severe hypotension that required pressor or surgery; Minor bleeding that required medical intervention to stop or treat bleeding: Minimal bleeding: any bleeding that did not require intervention or treatment such as bruising, bleeding gums, oozing from injection sites.

SECONDARY OUTCOMES:
value of Modified Rankin Scale(mRS) at three months | 3 months
  rmRS Measures the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability; its value ranges from 0 to 6; the lower the score, the better the stroke outcome. A favorable stroke outcome is considered with mRS value equal to two or less.
rate of composite recurrent stroke, myocardial infarction, and death due to vascular events | 3 months
  Rates of new stroke, TIA, myocardial infarction, or death from vascular events within three months of treatment, the investigators will perform follow-ups of the patient during visits to the outpatient clinic and perform needed investigations such as brain imaging, Electrocardiography, arterial and venous duplex ultrasound imaging
rate of drug adverse effects | 3 months
  all side effects related to the medications of our study will be reported

CONTACTS AND LOCATIONS:
Overall Officials: mohamed G. Zeinhom, MD, Principal Investigator — neurology department kafr el-sheikh university
Locations (1):
- Kafr Elsheikh University Hospital, Kafr ash Shaykh, Egypt

IPD SHARING:
Plan to Share IPD: No
All the data that support the findings of this research will be available from the corresponding author M. Zeinhom upon reasonable request.

REFERENCES:
- [Result] Paciaroni M, Ince B, Hu B, Jeng JS, Kutluk K, Liu L, Lou M, Parfenov V, Wong KSL, Zamani B, Paek D, Min Han J, Del Aguila M, Girotra S. Benefits and Risks of Clopidogrel vs. Aspirin Monotherapy after Recent Ischemic Stroke: A Systematic Review and Meta-Analysis. Cardiovasc Ther. 2019 Dec 1;2019:1607181. doi: 10.1155/2019/1607181. eCollection 2019. PMID 31867054
- [Result] Meyer DM, Albright KC, Allison TA, Grotta JC. LOAD: a pilot study of the safety of loading of aspirin and clopidogrel in acute ischemic stroke and transient ischemic attack. J Stroke Cerebrovasc Dis. 2008 Jan-Feb;17(1):26-9. doi: 10.1016/j.jstrokecerebrovasdis.2007.09.006. PMID 18190818